CLINICAL TRIAL: NCT00797589
Title: Effect of Prime Solution on Fluid Balance After Open Heart Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: B. Braun Melsungen AG (Industry)
Responsible Party: Principal Investigator, Alexey Schramko, MD, PhD, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008-001225-34
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Valve Surgery; Coronary Artery Bypass Grafting
Keywords: aorta valve; mitral valve; coronary artery bypass grafting surgery; perfusion; priming
MeSH Terms: interventions — Ringer's Lactate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ringer lactate (Experimental): Crystalloid solution
  Interventions: Drug: Ringer lactate
- HES solution (Tetraspan®) (Experimental): Balanced colloid solution
  Interventions: Drug: HES

INTERVENTIONS:
Drug: HES — 20ml/kg as prime fluid
  Arms: HES solution (Tetraspan®)
Drug: Ringer lactate
  Arms: Ringer lactate

SUMMARY:
The use of Tetraspan® as prime solution can reduce fluid extravasation after perfusion versus Ringer acetate. Plasma-adapted HES-solutions produce also less acidosis.

DETAILED DESCRIPTION:
Fifty patients scheduled for elective primary and single cardiac surgery include in this prospective study. Patients with preoperative coagulation disorders, or renal or hepatic failure, are excluded.

Before admission to the operation theatre, the patients allocate in random order to receive one of the following solutions during the extracorporeal circulation:

1. Ringer-acetate solution
2. 6% HES solution (Tetraspan®) During the 1 postoperative day we register hemodynamic changes, fluid balance, fluid extravasation, plasma ion concentration, modified thromboelastography, and kidney function.

ELIGIBILITY:
Inclusion Criteria:

* Elective combined cardiac surgery

Exclusion Criteria:

* Liver failure
* Kidney failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
fluid balance | 1 postoperative day

CONTACTS AND LOCATIONS:
Overall Officials: Raili T Suojaranta-Ylinen, MD, PhD, Study Chair — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland